CLINICAL TRIAL: NCT04354142
Title: iSpy: A Pilot Randomized Control Trial of a Novel Carbohydrate Counting Smartphone App for Youth With Type 1 Diabetes
Brief Title: A Novel Carbohydrate Counting Smartphone App for Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Mark Palmert, Associate Chair of Pediatrics, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000054297
Record Dates: First submitted 2020-04-10; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iSpy (Experimental): In addition to usual care, participants in the intervention group will receive the iSpy intervention.
  Interventions: Device: iSpy
- Control (No Intervention): The control group participants will continue to use their usual method of carbohydrate counting for a 3-month period.

INTERVENTIONS:
Device: iSpy — iSpy is a novel healthcare application that hopes to address an important clinical need by facilitating carbohydrate counting using pictures or voice recognition. Proprietary algorithms adjust for portion size and identify hidden carbohydrates (such as in ketchup or other condiments) and quantify the amount of carbohydrates in a meal.
  Arms: iSpy

SUMMARY:
Type 1 Diabetes Mellitus (T1DM) is a common chronic disease of childhood. T1DM has substantial impact on quality of life (QOL), including burdensome dietary restrictions and the need to count carbohydrates in foods to safely dose insulin. Carbohydrate counting is challenging, inconvenient, and, if done wrong, can cause high or low blood glucose levels.

To address these challenges, iSpy, a novel smartphone application, was created to identify foods and determine their carbohydrate content using pictures or speech. This pilot study is to evaluate if using iSpy improves carbohydrate counting accuracy and efficiency. Pilot participants will have carbohydrate counting (accuracy and efficiency) and their overall QoL (with respect to carbohydrate counting) assessed at baseline and after 3-months.

The investigators hypothesize that using iSpy will make carbohydrate counting easier (by improving accuracy and efficiency) and enhance QoL for patients and/or their caregivers. If so, iSpy may help lessen the burden of living with T1DM.

DETAILED DESCRIPTION:
Nutrition is an integral component of management of many chronic diseases and of overall wellness. Helping individuals to understand what they are eating can empower them to better manage their diseases. For example, the growing number of youth living with Type 1 Diabetes Mellitus (T1DM) struggle with carbohydrate counting, an essential and daily aspect of their lives, because of required reliance on memorization and numeracy skills. Effective carbohydrate counting has been demonstrated to improve blood glucose control, while inaccurate carbohydrate counting results in more variable blood glucose. Concerns related to carbohydrate counting accuracy can also limit food choices, provoke anxiety, and decrease quality of life. Since there is no cure for T1DM, enhancing patients' ability to understand and apply carbohydrate counting is an important part in helping them manage their condition most effectively.

iSpy is a novel healthcare application that addresses an important clinical need by facilitating carbohydrate counting using pictures or voice recognition. Proprietary algorithms adjust for portion size and identify hidden carbohydrates (such as in ketchup or other condiments) and quantify the amount of carbohydrates in a meal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T1DM for ≥6 months;
* Completion of initial carbohydrate counting classes;
* Incorporating carbohydrate counting into treatment regimen;
* Having access to a smart phone and data plan;

Exclusion Criteria:

* Cognitive impairments or co-morbid physical or psychiatric condition (e.g. blindness, clinical depression, anxiety disorder) that might impact ability to use iSpy;
* Diagnosis of condition that affects dietary exposure (e.g. celiac disease);
* Participation in usability study;

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Carbohydrate (CHO) Counting Accuracy | 3 months
  Assessing CHO counting using 10 food items from all major food groups. For each group, a simple food (e.g. an apple) and complex food (e.g. food with 2+ components but base food from targeted group) is included. A Co-investigator, Registered Dietitian (RD)/Certified Diabetes Educator (CDE), selected 2 sets of 10 food items for the study visits (verified that both sets were similar difficulty).
  The net CHO value (true value) for each food will be based on the nutrition label, USDA Nutrient Database (Release 28), Canadian Nutrient File, or by RD/CDE.
  For each food, data will be obtained from all participants:
  • Estimated net CHO (in grams)
  And with the above data, the following will be calculated:
  * % of food for which subjects estimated the CHO content within (+/-) 10 grams of true value.
  * Change (%) in the above accuracy measure for counting at baseline versus 3-month follow-up visit in iSpy vs control groups.
Carbohydrate (CHO) Counting Efficiency (Time to count) | 3 months
  Assessing CHO counting using 10 food items from all major food groups. For each group, a simple food (e.g. an apple) and complex food (e.g. food with 2+ components but base food from targeted group) is included. A Co-investigator, Registered Dietitian (RD)/Certified Diabetes Educator (CDE), selected 2 sets of 10 food items for the study visits (verified that both sets were similar difficulty).
  The net CHO value (true value) for each food will be based on the nutrition label, USDA Nutrient Database (Release 28), Canadian Nutrient File, or by RD/CDE.
  For each food, data will be obtained from all participants:
  • Time required to estimate net CHO (in seconds)
  In order to calculate the following:
  • Change in the above time taken for counting at baseline versus 3-month follow-up visit in iSpy vs control groups.

SECONDARY OUTCOMES:
Change in Quality of Life: Self Care Inventory Questionnaire | 3 months
  Quality of Life questionnaires will be analyzed for any change from baseline to 3-month follow-up within both the intervention and control groups.
  The first questionnaire including:
  • Self Care Inventory: Scale from 1 (Never do it) to 5 (Always do this as recommended without fail);
Change in Quality of Life: Diabetes Questionnaire | 3 months
  Quality of Life questionnaires will be analyzed for any change from baseline to 3-month follow-up within both the intervention and control groups.
  The second questionnaire including:
  • Diabetes Family Responsibility Questionnaire: Selection of 1 of 3 statements best describing the way each task is handled in the family from 1 (Parent taking responsibility almost all of the time) 2 (Parent and Child sharing responsibility equally) to 3 (Child taking responsibility almost all of the time);
Change in Quality of Life: Quality of Life for Youth | 3 months
  Quality of Life questionnaires will be analyzed for any change from baseline to 3-month follow-up within both the intervention and control groups.
  The third questionnaire including:
  • Quality of Life for Youth: Scale from 0 (Never) to 4 (All the time);
Change in Quality of Life: Global Quality of Life | 3 months
  Quality of Life questionnaires will be analyzed for any change from baseline to 3-month follow-up within both the intervention and control groups.
  The last questionnaire including:
  • Global Quality of Life: Scale from 1 (No Change) to 7 (A great deal better);
Implementation outcomes: Accrual/Attrition Rates | 3 months
  • Criteria for implementation success will be based on the studies previously conducted by Co-Principal Investigator (JS): Participant accrual (total completed / total enrolled) and attrition rates (total dropouts / total enrolled). Success being defined as accrual rates >70% and attrition rates <15%;
Implementation outcomes: Engagement | 3 months
  • Levels of engagement will be assessed as follows:
  * Low: defined as less than 1 logged meal every 2 weeks
  * High: defined as greater than 1 logged meal every 2 weeks.
Implementation outcomes: Acceptability | 3 months
  • Acceptability: 7 item Acceptability e-Scale (AES) regarding level of acceptability from a scale of 1 (low) to 5 (high) of iSpy, with high acceptability being item mean score of 4 on AES. 2 additional qualitative items are included in AES and will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Palmert, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alfonsi JE, Choi EEY, Arshad T, Sammott SS, Pais V, Nguyen C, Maguire BR, Stinson JN, Palmert MR. Carbohydrate Counting App Using Image Recognition for Youth With Type 1 Diabetes: Pilot Randomized Control Trial. JMIR Mhealth Uhealth. 2020 Oct 28;8(10):e22074. doi: 10.2196/22074. PMID 33112249